CLINICAL TRIAL: NCT03491514
Title: Glycemic and Insulinemic Impact of a Test Granola 3 Versus a Control Granola
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1711
Record Dates: First submitted 2018-03-31; First posted 2018-04-09 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Glycemic Response; Insulinemic Response; Subjectvie Hunger

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Granola (Experimental): 51 g of Test Granola
  Interventions: Other: Test Granola
- Control Granola (Placebo Comparator): 54.1 Control Granola
  Interventions: Other: Control Granola

INTERVENTIONS:
Other: Test Granola — 51 g Test Granola
  Arms: Test Granola
Other: Control Granola — 54.1 Control Granola
  Arms: Control Granola

SUMMARY:
The objectives of this study are to examine the blood glucose and serum insulin response elicited by servings of Test Granola and Control Granola containing equal amounts of available carbohydrate over a 3 h time period. In addition, the subjective hunger response to these foods will be measured over 3 h.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females, 18-65 years of age, inclusive
* Body mass index (BMI) between 21.0 and 32.0 kg/m², inclusive, at screening (visit 1).
* No participation in a PepsiCo study at GI Labs for at least 6 months from signing the consent form or previously enrolled into a PepsiCo Granola RAG:SAG trial (PEP-1701, PEP-1710).
* No participation in any clinical trial for at least 30 days from signing the consent form.
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
* Fasting serum glucose <7.0mmol/L or capillary whole blood glucose <6.3mmol/L.
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Wolever, the president of GI Testing, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or major surgical event within 6 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Lactose intolerance.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at screening.
* Change in body weight of >3.5kg within 4 weeks of the screening visit.
* Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 5 d prior to each test visit.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
* Exposure to any investigational product within 30 d prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Incremental area under the blood glucose curve | 0-2 hours

SECONDARY OUTCOMES:
Incremental areas under the curve of blood glucose | 0-3 hours; 2-3 hours
Incremental areas under the curve of serum insulin | 0-3 hours; 2-3 hours, 0-2 hours
subjective hunger | 0-2 hours, 0-3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Glycemic Index Laboratories, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No